CLINICAL TRIAL: NCT03161353
Title: Chemotherapy-free Trastuzumab and Pertuzumab in HER2-positive (Human Epidermal Receptor) Breast Cancer: FDG-PET Response-adapted Strategy. The PHERGain Study
Brief Title: Chemotherapy-free Trastuzumab and Pertuzumab in HER2-positive Breast Cancer: FDG-PET Response-adapted Strategy.
Acronym: PHERGain
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP096; 2016-002676-27 (EudraCT Number)
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Docetaxel; Carboplatin; Letrozole; Tamoxifen

STUDY DESIGN:
Intervention Model Description: This randomized, open-label phase II study will assess the efficacy of the combination of trastuzumab and pertuzumab, ± endocrine therapy according to HR (hormone receptor) status, as exclusive neoadjuvant and adjuvant treatment in patients with HER2-positive breast cancer through a FDG-PET response-adapted strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A (Experimental): Cohorts A/B if there is no evidence of subclinic M1 assessed by 18F-FDG PET/CT at screening. Interventional: Perjeta+Herceptin+Carboplatin+Docetaxel (during 4 cycles):
  PET responders or not responders after surgery: Continue with Perjeta+Herceptin+ Endocrine therapy (tamoxifen or letrozole) during 12 cycles
  A sub-set of 42 patients (35 patients from cohort A and 7 patients from cohort B) from 5 sites in Spain are participating in the LINGain sub-study "Prospective evaluation of predictive/prognostic immunogenicity biomarkers for target therapy in HER2-positive early breast cancer within the PHERGain study".
  Interventions: Drug: Perjeta; Drug: Herceptin; Drug: Docetaxel; Drug: Carboplatin; Drug: Letrozole; Drug: Tamoxifen
- Cohort B (Experimental): Cohorts A/B if there is no evidence of subclinic M1 assessed by 18F-FDG PET/CT at screening. Interventional: Perjeta+Herceptin+Endocrine therapy (tamoxifen or letrozole) during 2 cycles.
  * PET responders: Perjeta+Herceptin+Endocrine therapy during 6 cycles. -Complete response: continue with Perjeta+Herceptin+ Endocrine therapy during 10 cycles -Non-complete response: Perjeta+Herceptin+ Carboplatin+ Docetaxel during 6 cycles and Perjeta+Herceptin+Endocrine therapy during 4 cycles.
  * PET non-responders: Perjeta+Herceptin+Carboplatin+Docetaxel during 6 cycles. Patients with or without complete response will continue with Perjeta+Herceptin+Endocrine therapy during 10 cycles.
  A sub-set of 42 patients (35 patients from cohort A and 7 patients from cohort B) from 5 sites in Spain are participating in the LINGain sub-study "Prospective evaluation of predictive/prognostic immunogenicity biomarkers for target therapy in HER2-positive early breast cancer within the PHERGain study".
  Interventions: Drug: Perjeta; Drug: Herceptin; Drug: Docetaxel; Drug: Carboplatin; Drug: Letrozole; Drug: Tamoxifen
- Cohort C (Experimental): cohorts C if there is evidence of subclinic M1 assessed by 18F-FDG PET/CT at screening Interventional: Perjeta+Herceptin+Carboplatin+Docetaxel during 6 cycles. Patients will continue with Perjeta+Herceptin+Endocrine therapy (tamoxifen or letrozole) after surgery or no surgery.
  Interventions: Drug: Perjeta; Drug: Herceptin; Drug: Docetaxel; Drug: Carboplatin; Drug: Letrozole; Drug: Tamoxifen

INTERVENTIONS:
Drug: Perjeta — All patients will receive Perjeta® as an IV infusion on Day 1 of the first treatment cycle as a loading dose of 840 mg, followed by 420 mg on Day 1 of each subsequent 3-week cycle. Perjeta® IV should be administered 60 minutes after the end of Herceptin® SC (subcutaneous) administration. An observation period of 30-60 minutes is recommended after each Perjeta® infusion.
  Other Names: Pertuzumab
Drug: Herceptin — All patients will receive a fixed dose of 600 mg, irrespective of the patient's weight, will be administered throughout the treatment phase. All doses of Herceptin® SC will be administered as an SC injection into the thigh by a trained health care professional over a period of 2-5 minutes. No loading dose is required with Herceptin® SC.
  Other Names: Trastuzumab
Drug: Docetaxel — Docetaxel will be administered in line with the respective product information and/or recognized clinical practice guidelines. It will be administered after Herceptin® SC, Perjeta® IV, and carboplatin
Drug: Carboplatin — Carboplatin will be administered in line with the respective product information and/or recognized clinical practice guidelines. It will be administered after Herceptin® SC and Perjeta® IV.
Drug: Letrozole — Postmenopausal women will receive letrozole 2.5 mg tablet orally once daily beginning on Day 1 and continuing through Day 21 of a 21-day cycle as neoadjuvant therapy.
Drug: Tamoxifen — Premenopausal women will receive tamoxifen 20 mg tablet orally once daily beginning on Day 1 and continuing through Day 21 of a 21-day cycle as neoadjuvant therapy.
  Male patients will receive tamoxifen 20 mg tablet orally once daily beginning on Day 1 and continuing through Day 21 of a 21-day cycle as neoadjuvant therapy.

SUMMARY:
The study assess the early metabolic effects of neoadjuvant treatment with trastuzumab and pertuzumab (± endocrine therapy) on the primary tumor and axillary lymph nodes and their predictive value for pathologic complete response (pCR) in the breast and axilla.

And also assess 3-year invasive disease-free survival (iDFS) in patients with HER2-positive (HER: human epidermal receptor) breast cancer treated with neoadjuvant trastuzumab and pertuzumab (± endocrine therapy) using a FDG-PET response-adapted strategy.

DETAILED DESCRIPTION:
Investigational Medicinal Products (IMPs) will be trastuzumab and pertuzumab, carboplatin, and docetaxel, as well as all endocrine therapy drugs to be administered according to HR status (hormone receptor). For cohort C, trastuzumab SC (subcutaneous) and pertuzumab IV will be IMPs until a maximum of 18 cycles.

Patients will be randomly assigned in a 1:4 ratio, with a randomization stratified by HR status to receive trastuzumab and pertuzumab with docetaxel and carboplatin (cohort A) or trastuzumab and pertuzumab ± endocrine therapy according to HR status (cohort B).

A F-FDG PET/CT will be performed at baseline (total body) and after 2 cycles of neoadjuvant therapy. Central review of F-FDG PET/CT will be mandatory. Patients allocated into cohort A will continue with the same treatment for a total of six cycles regardless of 18F-FDG PET/CT results. Patients enrolled into cohort B showing at least 40% reduction of the SUVmax of F-FDG PET/CT respect to baseline (PET responders) will continue with the same treatment for a total of 8 cycles. PET-non responders patients will also receive neoadjuvant chemotherapy based on six cycles of docetaxel and carboplatin concurrently with trastuzumab and pertuzumab for all cycles.

Following surgery, cohort B/PET responders patients who do not achieve a pCR will additionally receive six cycles of docetaxel and carboplatin concurrently with trastuzumab and pertuzumab for all cycles. Moreover, all patients from cohorts A/B must complete 18 cycles of trastuzumab and pertuzumab, along with adjuvant endocrine therapy and radiotherapy according to HR status (hormone receptor) and institutional practices, respectively.

An additional exploratory cohort (cohort C) will include patients with evidence of subclinic M1 at baseline 18F-FDG PET/CT, but not previously detected by routine clinical assessment. These patients will receive trastuzumab and pertuzumab with docetaxel and carboplatin for a total of six cycles. After first six cycles, these patients will receive trastuzumab and pertuzumab ± endocrine.therapy according to HR status for at least 12 additional cycles after surgery (only if surgery is performed). According to institutional practices, it will be allowed to continue treatment with trastuzumab and pertuzumab, along endocrine therapy on the basis of HR status, as maintenance therapy until disease progression or unacceptable toxicity.

A sub-set of 42 patients (35 patients from cohort A and 7 patients from cohort B) from 5 sites in Spain are participating in the LINGain sub-study "Prospective evaluation of predictive/prognostic immunogenicity biomarkers for target therapy in HER2-positive early breast cancer within the PHERGain study" : Hospital General de Valencia, Hospital Clínico Universitario de Valencia, IVO, Hospital La Fe and Hospital Arnau de Vilanova.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures.
2. Female or male patients ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Histologically proven invasive breast cancer.
5. Operable breast cancer (cT1-3 and/or cN0-2 tumors) (breast cancer TNM classification)
6. Tumor size larger than or equal to 1.5 centimeter (cm) in diameter by magnetic resonance imaging (MRI) or ultrasound with a significant 18F-FDG uptake defined as maximum standarized uptake value (SUVmax: maximum standarized uptake value) ≥1.5 x SUVmean (mean standarized uptake value) liver + 2 SD (standard deviation.

Multicentric/multifocal tumors will be allowed only if:

1. Histological confirmation of at least two lesions.
2. All tumors must be HER2-positive.
3. Largest lesion must be larger than or equal to 1.5 cm in diameter by MRI or ultrasound.

7)Centrally confirmed HER2-positive disease according to the 2018 American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) criteria.

8)Patient must have known estrogen receptor (ER) and progesterone receptor (PR) status locally determined prior to study entry.

Patient has adequate bone marrow, liver, and renal function:

9)Hematological: White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x109/L, and hemoglobin ≥ 10.0 g/dL (≥ 6.2 mmol/L).

10)Hepatic: total bilirubin ≤ institutional upper limit of normal (ULN) (except for Gilbert's syndrome); alkaline phosphatase (ALP) ≤ 2.5 times ULN; aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 times ULN.

11)Renal: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

12)Patient must be accessible for treatment and follow-up.

Exclusion Criteria:

1. Previous treatment with chemotherapy, anti-HER2 therapy, radiation therapy, or endocrine therapy for invasive breast cancer.
2. cT4 and/or cN3 tumors (TNM breast cancer classification)
3. Bilateral breast cancer.
4. Evidence of metastatic disease by routine clinical assessment chest x-ray, liver ultrasound, and bone scan; or computed tomography (CT) scan of thorax and abdomen and bone scan, except patients with subclinic M1 (metastases) at baseline only according to 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT) that will be allowed to be included into cohort C.
5. Known hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances.
6. History of other malignancy within the last five years prior to first dose of study drug administration, except for curatively treated basal and squamous cell carcinoma of the skin and/or in situ cervical carcinoma.
7. Left ventricular ejection fraction (LVEF) below 55% as determined by multiple-gated acquisition (MUGA) scan or echocardiography (ECHO).
8. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) despite adequate antihypertensive treatment.
9. Clinically significant cardiovascular disease [stroke, unstable angina pectoris, or documented myocardial infarction within six months prior to study entry; history of documented congestive heart failure (CHF) (New York Heart Association II-III-IV); symptomatic pericarditis; documented cardiomyopathy; ventricular arrythmias with the exception of benign premature ventricular contractions; conduction abnormality requiring a pacemaker; other arrhythmias not controlled with medication].
10. Active uncontrolled infection at the time of enrollment.
11. Current known infection with HIV, hepatitis B virus, or hepatitis C virus.
12. Patients with pulmonary disease requiring continuous oxygen therapy.
13. Previous history of bleeding diathesis.
14. Patient is currently receiving anti-coagulant therapy, chronic treatment with corticosteroids, or another immunosuppressive agent (standard premedication for chemotherapy and local applications are allowed).
15. Major surgical procedure or significant traumatic injury within 14 days prior to randomization or anticipation of need for major surgery within the course of the study treatment.
16. Patient has other concurrent severe and/or uncontrolled medical conditions that would, in the investigator´s judgment, contraindicate her participation in the clinical study.
17. Concurrent participation in other clinical trial, except other translational studies.
18. History of receiving any investigational treatment within 28 days prior to randomization.
19. Pregnant or breast-feeding women or patients not willing to apply highly effective contraception as defined in the protocol.

LINGain sub-study: The LINGAIN project intends to include a total of 126 blood samples from PHERGain trial, as follows:

105 from patients treated with trastuzumab and pertuzumab ± endocrine therapy (according to HR status); 21 from patients treated with trastuzumab and pertuzumab + carboplatin and docetaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of pCR | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  evaluate the rate of pCR as defined by the absence of invasive disease in the breast and axilla (ypT0/isN0) at the time of surgery achieved with the combination of trastuzumab and pertuzumab (± endocrine therapy) as exclusive neoadjuvant treatment in PET responders patients (cohort B/PET responders) [PET/CT positive predictive value (PPV) for a pCR among patients who are PET responders].
3-year iDFS rate | After 3 years (36 months)
  time from the first date of no disease (i.e., date of surgery) to invasive recurrence, new invasive disease, or death by any cause. Recurrence will be defined in accordance with the standardized efficacy endpoints (STEEP) criteria. The primary analysis will be to estimate 3-year iDFS rate in cohort B.

SECONDARY OUTCOMES:
pCR rates in the breast and axilla (ypTO/isN0) | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  pCR rates in the breast and axilla (ypT0/isN0) (cohort A; cohort B; cohorts A/B by PET responder status).
pCR rates in the breast (ypT0/is) | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  pCR rates in the breast (ypT0/is) (cohort A; cohort B; cohorts A/B by PET responder status).
RCB score (residual cancer burden) | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  RCB score (cohort A; cohort B; cohorts A/B by PET responder status).
pCR rates in the breast and axilla | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  pCR rates in the breast and axilla (ypT0/isN0) (cohort A; cohort B; cohorts A/B by PET responder status; HR status, HER2 status and tumor stage).
Rate of breast conserving surgery | After Cycle 6 or 8 (each cycle 21 days- After 4.2 or 5.6 months)
  Rate of breast conserving surgery (cohort A; cohort B; cohorts A/B by PET responder status).
18F-FDG PET/CT response rate (18F-FDG: 18F-fluorodeoxyglucose) | After cycle 2 (each cycle 21 days- After 42 days approximately)
  18F-FDG PET/CT response rate (according to the adapted EORTC criteria) (cohort A; cohort B).
Optimal 18F-FDG PET/CT cut-off for pCR | After cycle 2 (each cycle 21 days-After 42 days approximately)
  Optimal 18F-FDG PET/CT cut-off for pCR (cohort A; cohort B).
Other 18FDG PET quantification parameters | After cycle 2 (each cycle 21 days- After 42 days approximately)
  Other 18F-FDG PET quantification parameters beside SUVmax for pCR (cohort A; cohort B). We will consider alternative measures to SUVmax in order to improve the ability to predict pCR; The best predictive parameter will be selected by means of logistic regressions models. For all tests, we will use two sided p-values with alpha ≤ 0.05 level of significance. The p-values emerging from these analyses will not be interpreted in a confirmative sense; they will be considered of descriptive nature only.
MRI response rate | After two cycles of neoadjuvant therapy, and prior to surgery (each cycle 21 days)
  MRI response rate (according to the RECIST criteria version 1.1) (cohort A; cohort B; cohorts A/B by PET responder status).
Health-related quality of life | Baseline, cycle 3 (after 63 days approximately), before surgery and end of study through study completion (after cycle 18- after 12 months approximately)
  Health-related quality of life (EORTC QLQ-C30- quality of life questionnaire and EORTC QLQ-BR23 quality of life questionnaires) (cohort A; cohort B; cohort C; cohorts A/B by PET responder status). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/quality of life scale, and six single itemsThe QLQ-BR23 (quality of life questionnaire) breast cancer module is meant for use among patients varying in disease stage and treatment modality.The scoring approach for the QLQ-BR23 (quality of life questionnaire) is identical in principle to that for the function and symptom scales/single items of the QLQ-C30.
3, 5, and 7-year iDFS | After 3, 5 and 7 years (After 36, 60 and 80 months)
  3, 5, and 7-year iDFS (cohort A; cohort B [with the exception of 3-year iDFS]; cohorts A/B by PET responder status, HR status, and HER2 status).
3,5 and 7-year DDFS (DDFS:Distant disease-free survival) | After 3, 5 and 7 years (After 36, 60 and 80 months)
  3, 5, and 7-year DDFS (cohort A; cohort B; cohorts A/B by PET responder status, HR status, and HER2 status).
3, 5 and 7-year DFS (DFS:Disease-free survival) | After 3, 5 and 7 years (After 36, 60 and 80 months)
  3, 5, and 7-year DFS (cohort A; cohort B; cohorts A/B by PET responder status, HR status, and HER2 status).
3, 5 and 7-year (OS: overall survival) | After 3, 5 and 7 years (After 36, 60 and 80 months)
  3, 5, and 7-year OS (cohort A; cohort B; cohort C; cohorts A/B by PET responder status, HR status, and HER2 status)
PFS (cohort C) (PFS: Progression-free survival) | Until progression or death, assessed up to approximately 84 months
  PFS (patients with subclinical M1 at baseline by 18F-FDG PET/CT - cohort C).
Adverse events | Until progression or death, assessed up to approximately 84 months
  Adverse events, grade 3-4 adverse events, related adverse events, serious adverse events, related serious adverse events, and adverse events leading to discontinuation (cohort A; cohort B; cohort C; cohorts A/B by PET responder status, HR status, and HER2 status).
3, 5, and 7-year EFS | After 3, 5 and 7 years (After 36, 60 and 80 months)
  3, 5, and 7-year EFS (cohort A; cohort B).
To assess 3, 5, and 7-year adapted iDFS, DDFS, and DFS | After 3, 5 and 7 years (After 36, 60 and 80 months)
  To assess 3, 5, and 7-year adapted iDFS, DDFS, and DFS on patients with subclinical M1 at baseline by 18F-FDG PET/CT - cohort C.

OTHER OUTCOMES:
LINGain sub-study: analyze the variation of peripheral γδ T cells in blood samples | Screening, end of cycle 1 and end of cycle 2 (each cycle is 21 days)
  To analyse the variation of peripheral γδ T cells in blood samples from patients with HER2-positive early breast cancer in neoadjuvant treatment with trastuzumab and pertuzumab (± endocrine therapy) at 6 weeks after start of treatment (end of the 2nd cycle of treatment) respect to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, MD, Principal Investigator — Hospital Arnau de Vilanova
Locations (56):
- Institute Jules Bordet, Brussels, Belgium
- France (7):
  - CLCC d'Auvergne. Centre Jean Perrin., Clermont-Ferrand
  - Institute de Cancerologie de Laurraine, Nancy
  - Groupe Hospitalier Diaconesses, Paris
  - Hopital Tenon, Paris
  - Hospital Georges Pompidou, Paris
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Régaud, Toulouse
- Germany (6):
  - Kliniken Essen Mitte, Essen
  - Klinikum der Med. Fakultät Halle, Halle
  - National center for tumor disease NCT, Heidelberg
  - Städtisches Klinikum "St. Georg" Leipzig, Leipzig
  - Clinical of Nuclear Medicine Technical University Munich, Munich
  - Hämatologisch-Onkologische Schwerpunktpraxis, München
- Italy (7):
  - Ospedale Maggiore Bologna, Bologna
  - Ospedale Antonio Perrino, Brindisi
  - Istituto Ospedalieri di Cremona, Cremona
  - Ospedale Mantova, Mantova
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo, Monza
  - Ospedale Guglielmo de Saliceto, Piacenza
- Portugal (7):
  - Hospital Senhora da Oliveira, Guimarães
  - Hospital Beatriz Angelo, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital Fernando Fonseca, Lisbon
  - Centro Hospitalar Sao Joao, Porto
  - Hospital do Santo Antonio, Porto
  - Centro Hospitalaer de Tras-os-Montes e Alto Douro, Vila Real
- Spain (25):
  - ICO Badalona, Badalona, Barcelona
  - ICO l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Provincial de Castellón, Castelló, Castelló
  - Hospital de Jaén, Jaén, Jaén
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital San Joan de Reus, Reus, Tarragona
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Vall D'Hebrón, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Reina Sofía, Córdoba
  - ICO Girona, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital La Paz, Madrid
  - Hospital Ramón y Cajal, Madrid
  - CHUS Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínic Universitari de Valencia, Valencia
  - Hospital Dr Peset, Valencia
  - Hospital General Universitari de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Universitario Miquel Servet, Zaragoza
- United Kingdom (3):
  - Barts Cancer Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Llombart-Cussac A, Prat A, Perez-Garcia JM, Mateos J, Pascual T, Escriva-de-Romani S, Stradella A, Ruiz-Borrego M, de Las Heras BB, Keyaerts M, Galvan P, Braso-Maristany F, Garcia-Mosquera JJ, Guiot T, Gion M, Sampayo-Cordero M, Di Cosimo S, Perez-Escuredo J, de Frutos MA, Cortes J, Gebhart G. Clinicopathological and molecular predictors of [18F]FDG-PET disease detection in HER2-positive early breast cancer: RESPONSE, a substudy of the randomized PHERGain trial. Eur J Nucl Med Mol Imaging. 2024 Jul;51(9):2733-2743. doi: 10.1007/s00259-024-06683-0. Epub 2024 Apr 8. PMID 38587643
- [Derived] Perez-Garcia JM, Cortes J, Ruiz-Borrego M, Colleoni M, Stradella A, Bermejo B, Dalenc F, Escriva-de-Romani S, Calvo Martinez L, Ribelles N, Marme F, Cortes A, Albacar C, Gebhart G, Prat A, Kerrou K, Schmid P, Braga S, Di Cosimo S, Gion M, Antonarelli G, Popa C, Szostak E, Alcala-Lopez D, Gener P, Rodriguez-Morato J, Mina L, Sampayo-Cordero M, Llombart-Cussac A; PHERGain Trial Investigators. 3-year invasive disease-free survival with chemotherapy de-escalation using an 18F-FDG-PET-based, pathological complete response-adapted strategy in HER2-positive early breast cancer (PHERGain): a randomised, open-label, phase 2 trial. Lancet. 2024 Apr 27;403(10437):1649-1659. doi: 10.1016/S0140-6736(24)00054-0. Epub 2024 Apr 3. PMID 38582092
- [Derived] Perez-Garcia JM, Gebhart G, Borrego MR, Schmid P, Marme F, Prat A, Dalenc F, Kerrou K, Colleoni M, Braga S, Malfettone A, Sampayo-Cordero M, Cortes J, Llombart-Cussac A. Trastuzumab and pertuzumab without chemotherapy in early-stage HER2+ breast cancer: a plain language summary of the PHERGain study. Future Oncol. 2022 Oct;18(33):3677-3688. doi: 10.2217/fon-2022-0663. Epub 2022 Oct 27. PMID 36300423
- [Derived] Perez-Garcia JM, Gebhart G, Ruiz Borrego M, Stradella A, Bermejo B, Schmid P, Marme F, Escriva-de-Romani S, Calvo L, Ribelles N, Martinez N, Albacar C, Prat A, Dalenc F, Kerrou K, Colleoni M, Afonso N, Di Cosimo S, Sampayo-Cordero M, Malfettone A, Cortes J, Llombart-Cussac A; PHERGain steering committee and trial investigators. Chemotherapy de-escalation using an 18F-FDG-PET-based pathological response-adapted strategy in patients with HER2-positive early breast cancer (PHERGain): a multicentre, randomised, open-label, non-comparative, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):858-871. doi: 10.1016/S1470-2045(21)00122-4. Epub 2021 May 18. PMID 34019819